CLINICAL TRIAL: NCT04830540
Title: Impact of 'Recovery' Footwear on Lower Extremity Comfort and Biomechanics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1826
Record Dates: First submitted 2021-03-05; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-02

CONDITIONS: Arthralgia; Joint Stiffness; Gait Mechanics
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants assigned to the control group will be asked to continue wearing their typical shoes and to complete every two weeks the footwear and injury log provided
- Intervention (Experimental): Individuals assigned to the intervention group will be provided with 2 styles of the OOFOS recovery shoes, and will be asked to wear the OOFOS slide, sandal and/or closed toe shoes as their primary footwear outside training and competition for the 6 weeks between study visits. Intervention participants will also be asked to complete a daily shoe wear log and a shoe comfort assessment survey every other week.
  Interventions: Device: OOFOS Recovery Footwear

INTERVENTIONS:
Device: OOFOS Recovery Footwear — The OOFOS shoes/ sandals are a commercially available footwear with a compliant, energy absorbing midsole material.
  Arms: Intervention

SUMMARY:
The goal of this study is to understand the impact of wearing shoes with a compliant, energy absorbing midsole material, outside of athletic training sessions on the mechanics of movement, performance, and perceived joint pain and stiffness. Advances in material science have led to a wider range of cushioning system material properties and mid and outsole geometries in footwear. While there are many marketing claims about the potential health benefits of this new class of footwear these have not yet been investigated in well-designed scientific studies.

It is hypothesized that the intervention shoe as compared to the control will reduce self-reported joint pain and stiffness, improve ankle plantarflexion function and increase intersegmental foot motion during walking.

DETAILED DESCRIPTION:
Participants will be asked to make 2 visits, 6 weeks apart, to the Umass Biomechanics Lab in the Totman Building at UMass Amherst for gait analysis and biomechanical performance testing.

At the first study visit, participants will be randomly assigned to one of two groups. Participants assigned to the control group will be asked to continue wearing their typical shoes and to complete every two weeks the footwear and injury log provided. Individuals assigned to the intervention group will be provided with 2 styles of the OOFOS recovery shoes, and will be asked to wear the OOFOS slide, sandal and/or closed toe shoes as their primary footwear outside training and competition for the 6 weeks between study visits. Intervention participants will also be asked to complete a daily shoe wear log and a shoe comfort assessment survey every other week.

At each study visit, subjects will be asked to read and sign an Informed Consent Form, and will also be asked questions about their health, exercise, and injury history. To prepare for the data collection, participants will be asked to change into a pair of shorts and tight shirt that will be provided. Anatomic measurements will then be made with a measuring tape, and ankle flexibility will be assessed by manually moving the participant's ankle into the most flexed and most extended position.

Reflective markers will then be placed on subject's feet/shoes, legs, thighs, hips, shoulders, and arms to record 3-D limb kinematics. To place the markers, we will put little circles of double-sided tape on skin or clothing, with reflective balls on the outer side. The position of the reflective markers will be recorded by high-speed infrared cameras surrounding the data collection space. Subjects will also be instrumented with electromyography (EMG) sensors on the skin over muscles of the leg, to measure the activity of those muscles. Before placing the EMG sensors, a small patch of skin will be shaved to ensure the sensor stays in place and captures the signals needed.

Once markers have been placed, subjects will stand in the data collection space to record a standing calibration trial of the markers. The standing calibration trial will be used to create a computer model on which data analysis will be performed. Subjects will then walk on a long walkway with the cameras surrounding it at a both self-selected and a set speed of 1.4 m/s. This will be repeated several times until at least 5 successful trials have been recorded. A successful trial means that the walking speed varies by no more than 5 % from the previous trial. Subjects will perform the walking trials barefoot and in the OOFOS sandal and closed toe shoes.

Following the gait analysis described above, calf muscle strength will be assessed using a dynamometer. The subject will sit with the leg, hips, and torso securely strapped to prevent unwanted movement. Subjects will then preform isometric and dynamic contractions; enough repetitions will be allowed to facilitate learning of the technique required.

The final test will be a maximum vertical jump height test. Subjects will stand in the middle of the motion capture area and jump as high as they can from a standing position.

When the above procedures are completed, the research staff will open the intervention assignment envelope that will determine if you are assigned to the intervention or control group.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 - 35 kg/m2.
* Stiff or cleated footwear athlete on a competitive team.

Exclusion Criteria:

* Current injury that required absence from one or more practices in the last 3 weeks of regular team practice.
* Orthotic or other shoe insert used outside of athletic training times.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Calf Muscles Strength | 2 - 3 hours on week 1
  Unilateral isometric and isokinetic strength based on maximal contractions performed on a dynamometer.
Calf Muscles Strength | 2 - 3 hours on week 6.
  Unilateral isometric and isokinetic strength based on maximal contractions performed on a dynamometer.
Gait Mechanics | Gait analysis test at week 1 with 5 trials of overground walking at a speed of 1.4 m/s
  Gait kinematics during overground walk at preferred speed, and 1.4m/s, evaluated with a motion capture system.
Gait Mechanics | Gait analysis test at week 6 with 5 trials of overground walking at a speed of 1.4 m/s
  Gait kinematics during overground walk at preferred speed, and 1.4m/s, evaluated with a motion capture system.
Muscle EMG activity | Gait analysis test at week 1 with 5 trials of overground walking at a speed of 1.4 m/s
  Unilateral Surface Electromyography of Medial Gastrocnemius, Lateral Gastrocnemius, Vastus Medialis, Vastus Lateralis, Tibialis Anterior, Peroneus Longus, Soleus, Biceps Femoris, and Semitendinosus, during overground walk.
Muscle EMG activity | Gait analysis test at week 6 with 5 trials of overground walking at a speed of 1.4 m/s
  Unilateral Surface Electromyography of Medial Gastrocnemius, Lateral Gastrocnemius, Vastus Medialis, Vastus Lateralis, Tibialis Anterior, Peroneus Longus, Soleus, Biceps Femoris, and Semitendinosus, during overground walk.
Maximum Vertical Jump | 2 - 3 hours on week 1
  Height (m) of center of mass above ground measured by markers place on posterior superior iliac spine.
Maximum Vertical Jump | 2 - 3 hours on week 6
  Height (m) of center of mass above ground measured by markers place on posterior superior iliac spine.
Self-reported shoe comfort | Week 0, 5 minutes
  Shoe wear and comfort log
Self-reported pain, and injury. | Week 0, 5 minutes
  Injury and pain log
Self-reported shoe comfort | Week 2, 5 minutes
  Shoe wear and comfort log
Self-reported pain, and injury. | Week 2, 5 minutes
  Injury and pain log
Self-reported shoe comfort | Week 4, 5 minutes
  Shoe wear and comfort log
Self-reported pain, and injury. | Week 4, 5 minutes
  Injury and pain log
Self-reported shoe comfort | Week 6, 5 minutes
  Shoe wear and comfort log
Self-reported pain, and injury. | Week 6, 5 minutes
  Injury and pain log

CONTACTS AND LOCATIONS:
Locations (1):
- Musculoskeletal & Orthopedic Biomechanics Laboratory/ University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No